CLINICAL TRIAL: NCT04769713
Title: Prospective Randomized Double-Blind Study of Pain Control With Hepatic Hilum Nerve Block Versus Sham Procedure For Hepatic Chemoembolization or Radiofrequency Ablation
Brief Title: Hepatic Hilar Nerve Block Versus Sham in Pain Control During Liver Ablation and TACE Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Louis-martin Boucher, Assistant Professor Diagnostic Radiology - Interventional Radiology Division, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-7139
Record Dates: First submitted 2020-12-08; First posted 2021-02-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pain Control; Liver Cancer
MeSH Terms: conditions — Agnosia; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Double-Blinded Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A technologist will either load up a syringe with ropivacaine or with saline. He will be the only one knowing what was put in the syringe. The operator will inject the content of the syringe at the location of the hepatic hilar nerve block, not knowing what is being injected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hepatic hilar nerve block in ablation patients (Experimental): 15ml of 0.7% ropivacaine will be injected at the hepatic hilum anterior to the portal vein as close to the bifurcation as possible under US guidance using a 21g needle prior to the Ablation procedure.
  Interventions: Procedure: Hepatic Hilar Nerve Block Needle placement; Drug: Injection of Ropivacaine in the hepatic hilum for the hepatic hilar nerve block
- Placebo procedure in ablation patients (Placebo Comparator): 15ml of sterile normal saline will be injected at the hepatic hilum anterior to the portal vein as close to the bifurcation as possible under US guidance using a 21g needle prior to the Ablation procedure.
  Interventions: Procedure: Hepatic Hilar Nerve Block Needle placement; Drug: Injection of normal saline in the hepatic hilum for the sham procedure
- Hepatic hilar nerve block in chemoembolization patients (Experimental): 15ml of 0.7% ropivacaine will be injected at the hepatic hilum anterior to the portal vein as close to the bifurcation as possible under US guidance using a 21g needle prior to the chemoembolization procedure.
  Interventions: Procedure: Hepatic Hilar Nerve Block Needle placement; Drug: Injection of Ropivacaine in the hepatic hilum for the hepatic hilar nerve block
- Placebo procedure in chemoembolization patients (Placebo Comparator): 15ml of sterile normal saline will be injected at the hepatic hilum anterior to the portal vein as close to the bifurcation as possible under US guidance using a 21g needle prior to the chemoembolization procedure.
  Interventions: Procedure: Hepatic Hilar Nerve Block Needle placement; Drug: Injection of normal saline in the hepatic hilum for the sham procedure

INTERVENTIONS:
Procedure: Hepatic Hilar Nerve Block Needle placement — Placement of a needle within 2cm of the portal vein bifurcation along its anterior surface for injection of nerve block agent (for nerve block) or saline (placebo) under US or CT guidance.
Drug: Injection of Ropivacaine in the hepatic hilum for the hepatic hilar nerve block — Injection of 15 ml 0.5% Ropivacaine at the hepatic hilum along the anterior surface of the portal vein within 2cm of the bifurcation.
  Arms: Hepatic hilar nerve block in ablation patients; Hepatic hilar nerve block in chemoembolization patients
Drug: Injection of normal saline in the hepatic hilum for the sham procedure — 15 ml sterile normal saline is injected at the hepatic hilum along the anterior surface of the portal vein within 2cm of the bifurcation.
  Arms: Placebo procedure in ablation patients; Placebo procedure in chemoembolization patients

SUMMARY:
This study is aimed at assessing the effectiveness of a novel liver specific nerve block in improving pain control during painful liver interventional radiology procedures including liver tumoral ablation and trans arterial chemoembolization, two procedures aimed at controlling liver tumors, but that can be associated with significant pain. This novel hepatic specific nerve block was designed by us and initial retrospective results suggests it might help in controlling such liver procedural derived pain. The study was designed to compare the liver block to a sham procedure in a blinded context and to follow the participants over three days post-procedure to asses for pain levels.

DETAILED DESCRIPTION:
This is a prospective study. Experienced interventional radiologists in the two McGill University Health Centre study centers (Royal Victoria Hospital and Montreal General Hospital) will perform all procedures:

* 80 consecutive subjects meeting the eligibility criteria, scheduled for chemoembolization of the liver for primary or secondary liver malignancies OR radiofrequency ablation of the liver for primary or secondary liver malignancies.
* Consent will be obtained from all patients by an interventional radiologist.
* All procedures will be performed by a qualified interventional radiology medical doctor (IRMD).
* Patients who accept to participate and fit the criteria will be randomized to either receive hepatic plexus block or a placebo control procedure, consisting of injection of normal saline.
* Hepatic hilum plexus nerve block will consist of the ultrasound-guided injection of ropivacaine at the hepatic hilum anterior to the portal vein as close to the bifurcation as possible. In the sham control group, the same location will be targeted, but only normal saline will be injected.
* A member of the radiology technologists will load the syringe with either ropivacaine or normal saline and the IRMD will thus be blinded to the patient's allocated group.
* All patients will be offered IV analgesia using midazolam and fentanyl during the procedure at set regular intervals as per our standard regimen.
* Similar IV analgesics as well as oral analgesics will be provided as per set orders during the recovery period in the post-procedural recovery room (PACU)
* The patient will be discharged home with standard prescriptions for home analgesics which include routine medication and medication to be used for breakthrough pain. While at home they will be entering pain surveys three times per day for three days.
* Data will be gathered, stored, and analyzed. The analysis will be stratified into patients who have received chemoembolization and patients who have received radiofrequency ablation.
* Follow-up of the patient will occur as per routine 4-6 weeks post chemoembolization/radiofrequency ablation to assess the clinical success of the therapeutic procedure (ablation and TACE) and patient satisfaction with pain control.

Subject data collection on the day of the procedure will include demographics, relevant medical history, vital signs before and during the procedure, use of IV analgesics, use of oral analgesics, use of nerve block or sham procedure and visual analogue pain scales at set intervals during hospital stay. Subject data collection while at home will include visual analogue pain scale and self-recording of medication intake.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to the Interventional Radiology department and approved for a chemo-embolization or radiofrequency ablation of malignant primary or secondary liver tumour.
2. At least 18 y.o.

Exclusion Criteria:

1. Patients in whom the vascular anatomy prevents safe access to the hepatic hilum or patients in whom general anaesthesia was performed.
2. Patients who have known allergy to any anaesthetic agent in the regular protocol (fentanyl, midazolam, ropivacaine).
3. Patients with signs of skin infection at the entry site of the needle used to perform the nerve block
4. Patients with signs of infection such as fever or acute increase in wight blood cell count.
5. Patients with uncorrectable abnormal coagulation status (INR >1.5 and platelets < 50000 without use of anticoagulation agents).
6. Patients with pre-existing conditions, which, in the opinion of the investigator, interfere with the conduct of the study (these reasons will be recorded)
7. Patients, who are uncooperative, cannot follow instructions, or who are unlikely to comply with follow-up appointments or fill-out the post-procedural pain questionnaires.
8. Patients with a mental state that may preclude completion of the study procedure or are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in pain after a hepatic hilar nerve block during and immediately after liver ablation | 1 day
  Visual analog pain score will be compared between patient having received the hepatic hilar nerve block versus those having had a placebo procedure done during the ablation procedure and while in post-anesthetic care unit. Visual analog scales are on a scale of 0-10 with 0 being no pain and 10 the worse pain imaginable.
Changes in narcotic use after a hepatic hilar nerve block during and immediately after liver ablation | 1 day
  Number of mg of narcotics used to control the pain during and immediately after the ablation while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo
Changes in pain after a hepatic hilar nerve block during and immediately after liver chemoembolization | 1 day
  Visual analog pain score will be compared between patient having received the hepatic hilar nerve block versus those having had a placebo procedure done during the chemoembolization procedure and while in post-anesthetic care unit. Visual analog scales are on a scale of 0-10 with 0 being no pain and 10 the worse pain imaginable.
Changes in narcotic use after a hepatic hilar nerve block during and immediately after liver chemoembolization | 1 day
  Number of mg of narcotics used to control the pain during and immediately after the chemoembolization while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo

SECONDARY OUTCOMES:
Changes in pain after a hepatic hilar nerve block in the early days following liver ablation | 3 days
  Visual analog pain score will be compared between patient having received the hepatic hilar nerve block versus those having had a placebo procedure done up to 3 days post ablation. Visual analog scales are on a scale of 0-10 with 0 being no pain and 10 the worse pain imaginable.
Changes in narcotic use after a hepatic hilar nerve block in the early days after liver ablation | 3 days
  Number of mg of narcotics used to control the pain in the next 3 days after the ablation while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo
Changes in pain after a hepatic hilar nerve block in the early days following liver chemoembolization | 3 days
  Visual analog pain score will be compared between patient having received the hepatic hilar nerve block versus those having had a placebo procedure done up to 3 days post chemoembolization. Visual analog scales are on a scale of 0-10 with 0 being no pain and 10 the worse pain imaginable.
Changes in narcotic use after a hepatic hilar nerve block in the early days after liver chemoembolization | 3 days
  Number of mg of narcotics used to control the pain in the next 3 days after the chemoembolization while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo
Changes in anti-nausea medication use after a hepatic hilar nerve block during and immediately after liver ablation | 1 day
  Number of mg of anti-nausea medication used to control the pain during and immediately after the ablation while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo
Changes in anti-nausea medication use after a hepatic hilar nerve block during and immediately after liver chemoembolization | 1 day
  Number of mg of anti-nausea medication used to control the pain during and immediately after the chemoembolization while in post-anesthetic care unit will be compared between the group having had the hepatic hilar nerve block and those having had the placebo
Incidence of complications secondary to performing the hepatic hilar nerve block | 4-6 weeks
  Incidence of complications (graded based on society of interventional radiology complication grading system) will be calculated for the various grades
Differences in disease response post liver tumoral ablation between patients with hepatic hilar nerve block and those with sham procedure | 4-6 weeks
  RECIST criteria scoring system will be used to compare treatment response on CT/MRI 4-6 weeks post liver tumoral ablation in patients having had the hepatic hilar block versus those having had the sham procedure
Differences in disease response post liver tumoral chemoembolization between patients with hepatic hilar nerve block and those with sham procedure | 4-6 weeks
  RECIST criteria scoring system will be used to compare treatment response on CT/MRI 4-6 weeks post liver tumoral chemoembolization in patients having had the hepatic hilar block versus those having had the sham procedure

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data